CLINICAL TRIAL: NCT06856395
Title: Effect of Using Educational Robots During Vaccination on Fear and Pain in Children
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Balikesir University (Other)
Responsible Party: Principal Investigator, Sibel Ergün, professor, Balikesir University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 0000-0003-1227-5856
Record Dates: First submitted 2025-02-15; First posted 2025-03-04 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Fear; Fear of Pain; Pain; Vaccination; Child Behavior
Keywords: pain; fear; vaccination; child behavior
MeSH Terms: conditions — Pain; Child Behavior

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial with 2 groups
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): The child patients in this group will be given the opportunity to get to know, touch and examine the educational mini robot for 5 minutes before the DaBT-İPA vaccination. The robot will attract the child's attention. During this time, the sociodemographic data form will be filled. At the end of the 5th minute, the child patient will be prepared for the vaccination with the cooperation of the staff and parents. During this time, the researcher will maintain the child's relationship with the robot and ensure that he/she focuses his/her attention on the robot. The application will end after the DaBT-İPA vaccination procedure. 5 minutes after the procedure, the Child Fear Scale (ÇKÖ, Wong Baker Pain Scale) will be filled by the researcher using the face-to-face interview technique. The robot will be cleaned with antiseptic solution after each child patient.
  Interventions: Other: intervention group
- control group (No Intervention): After the procedure is explained according to the child's developmental level, the DaBT-IPA vaccine will be administered in accordance with the institution's policies. After 5 minutes, the Sociodemographic data form, Child Fear Scale (CHS), Wong Baker Pain Scale will be filled out by the researcher using the face-to-face interview technique. At the end of the data collection, the control group will be provided with time to spend with the robot in order to be beneficial.

INTERVENTIONS:
Other: intervention group — Robotic distraction during vaccination process
  Arms: intervention group

SUMMARY:
Pain and fear are very common in children during vaccination. We are planning to conduct a study to help children go through this process more comfortably. The aim is to examine whether the educational robot has an effect on pain and fear during vaccination in 4-year-old children in a randomized controlled manner.

DETAILED DESCRIPTION:
Data Collection Method:

A sample group of 74 people will be divided into two groups using www.randomizer.org using a simple randomization method.

Intervention group: The child patients in this group will be given the opportunity to get to know, touch and examine the educational mini robot for 5 minutes before the DaBT-IPA vaccination. The robot will attract the child's attention. During this time, the sociodemographic data form will be filled. At the end of the 5th minute, the child patient will prepare the vaccination with the cooperation of the staff and parents. During this time, the researcher will maintain the child's relationship with the robot and ensure that he/she focuses his/her attention on the robot. The application will end after the DaBT-IPA vaccination process. 5 minutes after the procedure, the Child Fear Scale (ÇKÖ, Wong Baker Pain Scale) will be filled by the researcher using a face-to-face interview technique. The robot will be cleaned with antiseptic solution after each child patient. Control Group: After the procedure is explained according to the child's developmental level, the DaBT-İPA vaccine will be administered in accordance with the institution's policies. 5 minutes later, the Sociodemographic data form, Child Fear Scale (ÇKÖ, Wong Baker Pain Scale) will be filled by the researcher using a face-to-face interview technique. At the end of the data collection, the control group will be provided with the opportunity to spend time with the robot in order to be beneficial.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the study
* The child must be 4 years old
* Must have come to a primary care center in Balıkesir city center
* DaBT-İPA vaccination must be administered
* Vastus Lateralis muscle must be used in vaccination

Exclusion Criteria:

* Not volunteering to participate in the study
* The child is not 4 years old
* He/she has not come to a family health center in Balıkesir city center
* DaBT-İPA vaccination is not applied
* Vastus Lateralis muscle will not be used in vaccination application

Ages: 48 Months to 60 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 74 (Estimated)
Dates: Start 2025-03-31 (Estimated); Primary Completion 2025-11-30 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Pain status of participants in the experimental group post vaccination | 6 months
  Average pain scale score of participants in the experimental group after vaccination. In the Wong Baker pain scale, the lowest value is expressed as 0 and the highest value is expressed as 5.
Pain status of participants in the control group post vaccination | 6 months
  Average pain scale score of participants in the control group after vaccination. In the Wong Baker pain scale, the lowest value is expressed as 0 and the highest value is expressed as 5.

SECONDARY OUTCOMES:
Fear status of participants in the experimental group post vaccination | 6 months
  Average children fear scale score of participants in the experimental group after vaccination.In the children's fear scale, the lowest value is expressed as 0 and the highest value is expressed as 4.
Children fear status of participants in the control group post vaccination | 6 months
  Average children fear scale score of participants in the control group after vaccination.In the children's fear scale, the lowest value is expressed as 0 and the highest value is expressed as 4.